CLINICAL TRIAL: NCT04407169
Title: Evaluation of the Prevalence of Critical Forms of CoVid-19 in Patients With Chronic Respiratory Disease Hospitalized for Severe Forms
Brief Title: Prevalence of Critical Forms of CoVid-19 in Patients With Chronic Respiratory Disease
Acronym: CRITICoVid
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI081
Record Dates: First submitted 2020-04-14; First posted 2020-05-29 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-05

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without chronic respiratory disease: All patients hospitalized for severe CoVid-19 without chronic respiratory disease
  Interventions: Other: no intervention
- Patients with chronic respiratory diseas: Patients hospitalized for severe CoVid-19 with one chronic respiratory disease
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — There will be no intervention. It is only an observationnal study

SUMMARY:
A new Coronavirus (SARS-CoV-2) emerged in Wuhan Province, China in December 2019 and rapidly spread around the world. To date, the data in the literature regarding the clinical and epidemiological characteristics of severe forms of CoVid-19 in patients with chronic respiratory disease are not well known.

The hypothesis is that patients with chronic respiratory disease (COPD, asthma, bronchial dilatations, pulmonary hypertension, cystic fibrosis, obesity-hypoventilation syndrome, obstructive sleep apnea syndrome) infected with SARS-Cov-2 will have increased dyspnea and hypoxemia leading to hospitalization for severe forms more frequently than the general population. However, they do not appear to be more at risk of developing a critical form.

This study is carried out in order to propose to estimate the prevalence of critical forms of CoVid19 among patients with chronic respiratory diseases hospitalized for severe forms.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* Diagnosis of CoVid-2 SARS infection retained (from clinical presentation, radiological and CoVid-19 positive microbiological specimen).
* Hospitalisation in the conventional medical sector for "respiratory" reasons (= severe form of CoVid-19) in the Nancy-Brabois hospital and Metz-Thionville Hospital between 02/03/2020 and 15/06/2020.

Exclusion Criteria:

* Diagnosis of SARS-CoV-2 infection not retained
* Refusal of the patient to participate in the study
* Persons referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code: o Pregnant woman, parturient or breastfeeding mother o Minors (not emancipated) o Persons of full age subject to a legal protection measure (guardianship, curatorship, safeguard of justice) - Persons of full age unable to express their consent Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care by virtue of articles L. 3212-1 and L. 3213-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized for severe CoVid-19 with or without chronic respiratory disease
Sampling Method: Probability Sample
Enrollment: 617 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who reached, during their hospitalization, a value greater than or equal to 6 on the WHO CoVid-19 infection progression scale | up to 28 days (during hospitalisation)
  Value of 6 or greeter on WHO CoVid-19 scale, indicating of a critical form of CoVid-19.

SECONDARY OUTCOMES:
Determined potential predictive factors of critic form in patients with chronic lung diseases | up to 28 days (during hospitalisation)
  Radiological damage (extension of ground-glass) could be a predictive factor.
Determined percentage of death | up to 28 days (during hospitalisation)
  intra-hospital death, intra-ICU death
Determined duration of oxygen therapy | up to 28 days (during hospitalisation)
  in days (or duration at a different flow rate compared to long-term home oxygen therapy prior to hospitalization)
Determined duration of hospitalization | up to 28 days (during hospitalisation)
  in days for patients with chronic respiratory disease between the date of admission and the date of discharge. Patients who died during hospitalization will be assigned the highest cohort value.
Determine mean values of the WHO CoVid-19 infection progression scale measured | up to 28 days (during hospitalisation)
  values will be measured at D3, D7 and D14 in each of the groups. Patients who do not reach D7 and D14 will have the last postponement

CONTACTS AND LOCATIONS:
Locations (1):
- Valentin Simon, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Fang L, Gao P, Bao H, Tang X, Wang B, Feng Y, Cong S, Juan J, Fan J, Lu K, Wang N, Hu Y, Wang L. Chronic obstructive pulmonary disease in China: a nationwide prevalence study. Lancet Respir Med. 2018 Jun;6(6):421-430. doi: 10.1016/S2213-2600(18)30103-6. Epub 2018 Apr 9. PMID 29650407
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Zhang JJ, Dong X, Cao YY, Yuan YD, Yang YB, Yan YQ, Akdis CA, Gao YD. Clinical characteristics of 140 patients infected with SARS-CoV-2 in Wuhan, China. Allergy. 2020 Jul;75(7):1730-1741. doi: 10.1111/all.14238. Epub 2020 Feb 27. PMID 32077115